CLINICAL TRIAL: NCT01783665
Title: The Effect of Aerobic Exercise on Cognitive Function and Sleep Quality in Individuals With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catherine Siengsukon, PT, PhD (Other)
Responsible Party: Sponsor-Investigator, Catherine Siengsukon, PT, PhD, Assistant Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13332
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2016-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Exercise (Experimental): 3x/week supervised moderate intensity aerobic exercise on recumbent stepper
  Interventions: Other: aerobic exercise
- Home exercise program (Active Comparator): Walking and stretching exercises performed 3x/week for 30 minutes at intensity considered non-aerobic
  Interventions: Other: home exercise program

INTERVENTIONS:
Other: aerobic exercise
  Arms: Aerobic Exercise
Other: home exercise program
  Arms: Home exercise program

SUMMARY:
In addition to the typical motor and sensory impairments, individuals with multiple sclerosis (MS) often experience cognitive dysfunction and sleep disturbances. Cognitive impairment occurs in 40 % - 70% of patients with MS. In addition, sleep problems in individuals with MS are very common, and approximately 50% of patients with MS have a diagnosable sleep disorder. The research believes that aerobic exercise improve cognitive function and improve sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of relapsing remitting or secondary progressive MS
* score 3-7 on the EDSS
* score < 55 on the Symbol Digit Modalities Test
* score > 5 on the Pittsburgh Sleep Quality Index

Exclusion Criteria:

* history of alcohol/drug abuse or nervous system disorder other than MS
* severe physical, neurological, or sensory impairments that would interfere significantly with testing
* developmental history of learning disability or attention-deficit/hyperactivity disorder
* relapse and/or corticosteroid use within four weeks of assessment
* unable to give consent
* uncorrected vision loss that would interfere significantly with testing
* score less than 24 on MMSE
* Acute ischemic cardiovascular event or coronary artery bypass surgery less than 3 months ago
* Either unable to physically perform the exercise test using the recumbent stepper or demonstrate absolute indications for terminating exercise that follows the American College of Sports Medicine's (ACSM) guidelines
* Uncontrolled blood pressure with medication (BP > 190/110mmHg)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Function | Baseline to Month 3

SECONDARY OUTCOMES:
Change in Sleep Quality | Baseline to Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Siengsukon, PT, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States